CLINICAL TRIAL: NCT03921450
Title: Overcoming Psychomotor Slowing in Psychosis (OCoPS-P): a 3-week, Randomized, Double-blind, Placebo-controlled Trial of add-on Repetitive Transcranial Magnetic Stimulation for Psychomotor Slowing in Psychosis
Brief Title: Overcoming Psychomotor Slowing in Psychosis (OCoPS-P)
Acronym: OCoPS-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-02164
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Schizophrenia and Related Disorders; Schizophrenia; Schizoaffective Disorder; Brief Psychotic Disorder
Keywords: motor behavior; psychomotor slowing; psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Motor Activity; Psychomotor Disorders

STUDY DESIGN:
Intervention Model Description: 3 week intervention with 15 sessions of add-on rTMS in 4 parallel arms, randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will not know the stimulation protocol, neither will the outcome assessor or the mental health care provider know the protocol applied
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Inhibitory repetitive transcranial magnetic stimulation (rTMS) (Experimental): 1 Hz stimulation of 17 mins over the supplementary motor area (SMA), 1000 pulses at 110% resting motor threshold intensity total of 15 sessions in 3 weeks
  Interventions: Device: 1 Hz rTMS
- Facilitatory intermittent theta burst stimulation (iTBS) (Active Comparator): Intermittent theta burst stimulation of 50 Hz over the supplementary motor area (SMA) with 600 pulses in 2 sec trains every 10 seconds for 190 seconds total. Two iTBS stimulations will be administered with 15 mins pause in between.
  total of 15 sessions in 3 weeks
  Interventions: Device: iTBS
- Placebo (Placebo Comparator): 1 Hz stimulation of 17 mins over the supplementary motor area (SMA) without any magnetic emission using a placebo-coil that looks identical and makes identical sounds as the real TMS coil total of 15 sessions in 3 weeks
  Interventions: Drug: Placebo
- Waiting group (No Intervention): This group will receive no intervention for 3 weeks. Afterwards they will receive the inhibitory rTMS protocol as in the first arm

INTERVENTIONS:
Device: 1 Hz rTMS — 1 Hz stimulation at 110% of resting motor threshold over supplementary motor area
  Arms: Inhibitory repetitive transcranial magnetic stimulation (rTMS)
Device: iTBS — 50 Hz theta burst stimulation at 80% of resting motor threshold over supplementary motor area
  Arms: Facilitatory intermittent theta burst stimulation (iTBS)
Drug: Placebo — 1 Hz stimulation with the placebo TMS coil without any magnetic emission
  Arms: Placebo

SUMMARY:
Psychomotor slowing is a major problem in psychosis. Aberrant function of the cerebral motor system is linked to psychomotor slowing in patients, particularly resting state hyperactivity in premotor cortices. A previous clinical trial indicated that inhibitory stimulation of the premotor cortex would reduce psychomotor slowing. The current study is further exploring this effect in a randomized, placebo-controlled, double-blind design with three arms of transcranial magnetic stimulation and measures of brain imaging and physiology prior to and after the intervention.

DETAILED DESCRIPTION:
As psychomotor slowing is a major problem in schizophrenia, contributing to poor functional outcome, and as no current treatment is effectively targeting psychomotor slowing, this study seeks to test noninvasive brain stimulation to overcome psychomotor slowing. Previous studies documented an aberrant increase of neural activity within the supplementary motor area (SMA) in patients with schizophrenia who had psychomotor slowing. Furthermore, a pilot study in major depression and schizophrenia indicated that inhibitory 1 Hz repetitive transcranial magnetic stimulation (rTMS) would improve psychomotor slowing in 82% of the participants. While this is encouraging, further evidence is needed to 1) replicate the clinical effect of 1 Hz rTMS on the SMA in schizophrenia, 2) to test against sham stimulation, facilitatory stimulation and no intervention, and 3) to test the effects of rTMS on the neural circuitry. Therefore, OCoPS includes more patients, more treatment arms, and more outcome variables than the first pilot trial.

Here we will enroll 88 patients with schizophrenia spectrum disorders and severe psychomotor slowing according to a standard rating scale. Subjects will be randomized to four arms, three of which are double blinded.

three weeks of daily rTMS over the SMA will be delivered. The first group receives inhibitory 1 Hz rTMS, the second group receives facilitatory intermittent theta burst stimulation (iTBS), and the third group receives sham stimulation with a placebo-coil. The fourth group will have no rTMS during the first three weeks, but will repeat the baseline measures after three weeks and then enter a treatment with 1Hz rTMS for three weeks. Outcome measures include the Salpetriere Retardation Rating Scale, observer ratings of motor behavior as well as measures of functioning. After the interventions, follow-up visits are planned at week 6 and week 24.

Finally, at baseline and after the rTMS course, patients will undergo MRI scanning for structural and functional alterations of the cerebral motor system.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed subjects
* Ability and willingness to participate in the study
* Ability to provide written informed consent
* Informed Consent as documented by signature
* Schizophrenia spectrum disorder according to diagnostic and statistical manual version 5 (DSM-5) criteria with current psychomotor slowing according to the Salpetriere Retardation Rating Scale (SRRS), score >= 15

Exclusion Criteria:

* Substance abuse or dependence other than nicotine
* Past or current medical or neurological condition associated with impaired or aberrant movement, such as brain tumors, stroke, M. Parkinson, M. Huntington, dystonia, or severe head trauma with subsequent loss of consciousness.
* Epilepsy or other convulsions
* History of any hearing problems or ringing in the ears
* Standard exclusion criteria for MRI scanning and TMS; e.g. metal implants, claustrophobia
* Patients only: any TMS treatment in the past 3 months
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Controls only: history of any psychiatric disorder or first-degree relatives with schizophrenia spectrum disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Proportion of responders at week 3 | Week 3
  Proportion of participants with >30% reduction from baseline in the Salpetriere Retardation Rating Scale (SRRS)
Change in Salpetriere Retardation Rating Scale (SSRS) from baseline | Week 3, week 6, week 24
  Change in the Salpetriere Retardation Rating Scale (SRRS) from baseline; the total score of 15 items is used, ranging 0-60 with higher scores indicating worse outcome

SECONDARY OUTCOMES:
Change in catatonia severity from baseline to week 3 | Week 3, week 6, week 24
  Observer based rating of catatonia severity with the Bush Francis Catatonia Rating Scale (BFCRS), assessment blind to intervention, total score of the BFCRS is used ranging 0-69 , with higher scores indicating poorer outcome
Change in negative symptoms from baseline | Week 3, week 6, week 24
  Change in the Brief Negative Symptom Scale (BNSS) from baseline, total score is used, ranging from 0-78 with higher values indicating poorer outcome, i.e. more negative symptom severity
Change in psychosis severity from baseline | Week 3, week 6, week 24
  Change in the Positive And Negative Symptom Scale (PANSS) from baseline, PANSS total score assesses the severity of positive, negative and general symptoms, ranging from 30-210 with higher scores indicating increased symptom severity, i.e. poorer outcome
Change in physical activity self report from baseline | Week 3, week 6, week 24
  Change in the International Physical Activity Questionnaire (IPAQ), the total score is used ranging from 0-70000 metabolic equivalent (MET)
Change in objectively measured physical activity from baseline | Week 3, week 6, week 24
  Change in the activity levels using wrist actigraphy
Change in dexterity from baseline | Week 3, week 6, week 24
  Change in the coin rotation task from baseline
Change in cortical excitability of the motor cortex from baseline | Week 3, week 6, week 24
  Change in Short Interval Cortical Inhibition (SICI) from baseline
Change in social and community functioning | Week 3, week 6, week 24
  Change in Social and Occupational Functional Assesment Scale (SOFAS) from baseline, the score ranges from 0-100 with higher scores indicating better functioning, i.e. better outcome
Change in functional capacity | Week 3, week 6, week 24
  Change in the Score of the brief version of the University of California, San Diego, Performance-Based Skills Assessment (UPSA-brief) assessment from baseline, higher scores indicating better function, the total score is used ranging 0-100
Change in functional connectivity | Week 3
  Change in the resting state functional connectivity within the cerebral motor system based on functional magnetic resonance imaging scans from baseline
Change in resting state cerebral perfusion | Week 3
  Change in the resting state cerebral perfusion within the cerebral motor system based on functional magnetic resonance imaging scans from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Walther, MD, Principal Investigator — University of Bern
Locations (1):
- University Hospital of Psychiatry, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walther S, Alexaki D, Weiss F, Baumann-Gama D, Kyrou A, Nuoffer MG, Wuthrich F, Lefebvre S, Nadesalingam N. Psychomotor Slowing in Psychosis and Inhibitory Repetitive Transcranial Magnetic Stimulation: A Randomized Clinical Trial. JAMA Psychiatry. 2024 Jun 1;81(6):563-571. doi: 10.1001/jamapsychiatry.2024.0026. PMID 38416468

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT03921450/Prot_SAP_000.pdf